CLINICAL TRIAL: NCT04914091
Title: Pilot Study for Quality Of Life and Drug Use Assessment in Patients With CAR-T Cells
Brief Title: Quality Of Life and Drug Use in Patients With CAR-T Cells
Acronym: QOLD CAR-T
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1182
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Patients With Diffuse Large B-cell Lymphoma Treated With CART-cells
Keywords: CAR-T cells; Quality of life; drug use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diffuse large B-cell lymphoma treated with CART-cells
  Interventions: Other: Semi-structured interviews and self-administered questionnaires

INTERVENTIONS:
Other: Semi-structured interviews and self-administered questionnaires — Interviews and questionnaires will be performed before administration of CAR-T cells, 3 month after and 6 month after, and will last 60 minutes each time. Semi-structured interview using pre-established questionnaires will be completed with a hospital pharmacist, concerning the patient's perception of his family, socio-professional environment, his knowledge of his illness and his treatment, the consumption of prescribed drugs outside the hospital, self-medication, complementary alternative therapies including herbal medicine. Seven self-administered questionnaires will be completed, concerning quality of life, Assessment of Cancer Treatment-Lymphoma, Beliefs about Medicines, Brief Illness Perception, satisfaction with medication, perceived social support scale, and on Health Literacy.

SUMMARY:
CAR-T cells are a major therapeutic innovation in the management of patients with relapsed or refractory diffuse large B cell lymphoma (DLBCL) in 3rd line or more. Kymriah® and Yescarta® are the first CAR-T with Marketing Authorization and coverage by the French Health Insurance. Their clinical interest has been demonstrated in non-comparative phase 1-2 trials.

The non-comparative design of the pivotal trials, the lack of data on patients' quality of life and drug consumption, as well as the very high cost of CAR-T (about € 320,000 for one treatment) warrant further studies.

This prospective non-comparative study aims to describe in real life the quality of life of patients treated with CAR-T cells, real world drug use and patients' experience feedback.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Eligible for treatment with CAR-T cells (outside any clinical trial) in an indication of DLBCL and for which treatment is scheduled
* Follow-up in the Hematology department of the Hospices Civils de Lyon
* Without major psychiatric disorder likely to interfere with the conduct of the study, in the opinion of the investigator
* Having given his non-opposition to participate in the study.

Exclusion Criteria:

* In an institution
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse large B-cell lymphoma treated with CART-cells in the center during the inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2033-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Mean quality of life score using the EORTC-QLQ C30 questionnaire | Inclusion (the day before lymphodepletion chemotherapy), Month 3 and Month 6 after the administration of CART-T cells
  Self-administered questionnaire EORTC-QLQ C30 (European Organisation for Research and Treatment of Cancer), developed to assess the quality of life of cancer patients, with 30 items. Score ranges from 0 (the worse) to 100 (the best).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon -Groupement Hospitalier Sud Service pharmaceutique, Unité de Pharmacie Clinique Oncologique, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No